CLINICAL TRIAL: NCT01140880
Title: Optimizing Access to Non-occupational Post Exposure Prophylaxis for HIV Using Contingency Management in Stimulant-Using Men Who Have Sex With Men
Brief Title: Biobehavioral Interventions for HIV-negative, Stimulant Using Men Who Have Sex With Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MC08-LA-710-FRI
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV Seroconversion; Stimulant Abuse
Keywords: Methamphetamine; Amphetamine; Cocaine; HIV; Post-exposure prophylaxis; HIV seronegativity
MeSH Terms: conditions — HIV Seropositivity | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contingency Management (Experimental): Participants will submit a urine sample every Monday, Wednesday, and Friday for 8 weeks (a total of 24 urine samples). Samples will be tested for stimulant metabolites. Increasingly valuable incentives will be provided for urine samples that lack metabolites of stimulant drugs.
  Participants reporting recent (i.e., < 48 hours) exposure to HIV viral inoculum will have the opportunity to initiate Truvada (1 pill daily for 28 days).
  Interventions: Drug: Truvada
- Yoked Contingency Management (Sham Comparator): Participants will submit a urine sample every Monday, Wednesday, and Friday for 8 weeks (a total of 24 urine samples). Samples will be tested for stimulant metabolites. Incentives will be provided to participants independent of stimulant drug use and determined in the same rate and timing as a randomly selected participant in the active CM condition.
  Participants reporting recent (i.e., < 48 hours) exposure to HIV viral inoculum will have the opportunity to initiate Truvada (1 pill daily for 28 days).
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Truvada At qualifying exposure, participants will take 28 days' worth (at one pill per day) of 200 mg emtricitabine and 300 mg tenofovir DF (Truvada).
  Other Names: Tenofovir/emtricitabine

SUMMARY:
This study seeks to evaluate the efficacy of a contingency management (CM) intervention compared to a yoked control condition for eliminating illicit stimulant use and for decreasing time to initiating post exposure prophylaxis (PEP), for improving adherence to PEP, and for completing PEP following a potential HIV-exposure event. Men who have sex with men who use cocaine amphetamine or methamphetamine frequently also have high risk sexual behaviors during or after their drug use. The objective of this study evaluates whether the use of CM that targets stimulant use significantly aids men who have sex with men who use stimulants and also engage in high-risk sexual transmission behaviors to be able to initiate, adhere to and complete PEP, thereby optimizing the utility of a biomedical HIV prevention intervention for reducing HIV incidence in this very high-risk group of MSM.

DETAILED DESCRIPTION:
This was a prospective, randomized study. 170 participants who met inclusion and exclusion criteria were randomized to CM or NCYC (non-contingent yoked-control condition) arms. They were provided with a 4-day starter-pack of PEP medication (tenofovir + emtricitabine, Truvada) to be started only in the event of a high-risk sexual exposure. The two interventions were implemented simultaneously:

The CM or NCYC intervention, remunerating (via vouchers) the participant based on his own (CM) or a yoked-participant's (NCYC) stimulant-metabolite-free urine samples for 8 weeks;

and,

Post-exposure prophylaxis, providing risk reduction counseling, adherence counseling and PEP medication for 28 days in the event of a high-risk sexual exposure to HIV.

All participants were followed for 24 weeks, or 24-weeks post-HIV-exposure, whichever was longer.

ELIGIBILITY:
Inclusion Criteria:

* Male who has sex with other men (MSM) by self-report
* At least 18 years of age
* HIV-negative serostatus on baseline rapid oral HIV antibody test, and no signs or symptoms consistent with primary HIV infection (PHI)
* Self-reported stimulant use within the previous 30 days
* Self-report of unprotected anal intercourse (either receptive or insertive) with an HIV-positive or status unknown partner within the previous 3 months
* Self-report of no previous hypersensitivity to any of the components of Truvada (tenofovir disoproxil fumarate or emtricitabine)
* In the opinion of the study medical provider, no contraindication to PEP medication treatment (laboratory testing, medical/drug interaction, or other)
* Has not used PEP in the previous 6 months
* A current resident of Los Angeles County
* Does not have a plan to move away from Los Angeles County in the next 6 months
* Willing and able to provide informed consent
* Willing and able to comply with study requirements

Exclusion Criteria:

* Does not identify as a male who has sex with other men
* Under 18 years of age
* HIV positive by self-report or as indicated by the results on baseline rapid oral HIV antibody testing
* Has not used a stimulant in the previous 30 days by self-report
* Has not had unprotected anal intercourse (either receptive or insertive) with an HIV-positive or status unknown partner within the previous 3 months
* Creatinine clearance <30 ml/min and not on dialysis
* Self-reports any previous hypersensitivity to any of the components of Truvada (tenofovir disoproxil fumarate or emtricitabine);
* In the opinion of the study medical provider, there exists a contraindication to administering Truvada-based post-exposure prophylaxis (laboratory testing, medical/drug interaction, or other)
* Has used PEP in the previous six months
* Not a current resident of Los Angeles County
* Unwilling or unable to provide informed consent
* Unwilling or unable to comply with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy J. Reback, Ph.D., Principal Investigator — Friends Research Institute, Inc.; Raphael J. Landovitz, M.D., M.Sc., Principal Investigator — UCLA Center for Clinical AIDS Research and Education; Steven Shoptaw, Ph.D., Principal Investigator — UCLA Department of Family Medicine
Locations (1):
- Friends Community Center, A Division of Friends Research Institute, Inc., Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Contingency Management: Participants will submit a urine sample every Monday, Wednesday, and Friday for 8 weeks (a total of 24 urine samples). Samples will be tested for stimulant metabolites. Increasingly valuable incentives will be provided for urine samples that lack metabolites of stimulant drugs.
  Truvada: Truvada At qualifying exposure, participants will take 28 days' worth (at one pill per day) of 200 mg emtricitabine and 300 mg tenofovir DF (Truvada).
- Yoked Contingency Management: Participants will submit a urine sample every Monday, Wednesday, and Friday for 8 weeks (a total of 24 urine samples). Samples will be tested for stimulant metabolites. Incentives will be provided to participants independent of stimulant drug use and determined in the same rate and timing as a randomly selected participant in the active CM condition.
  Truvada: Truvada At qualifying exposure, participants will take 28 days' worth (at one pill per day) of 200 mg emtricitabine and 300 mg tenofovir DF (Truvada).
Period: Overall Study
Arm/Group | Contingency Management | Yoked Contingency Management
Started | 70 | 100
Completed | 56 | 56
Not Completed | 14 | 44
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 8 | 10
Not completed — Protocol Violation | 0 | 30

BASELINE CHARACTERISTICS:
Population: 170 participants enrolled. 30 participants in the Yoked Contingency Management arm were involved in a protocol violation that rendered their data unusable. An additional 14 participants from each arm were either withdrawn, died (n = 1, not study related), or were lost to follow-up. Thus, baseline N = 140 (70/70), and follow-up N = 112 (56/56).
Groups:
- Total: Total of all reporting groups
Arm/Group | Contingency Management | Yoked Contingency Management | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.3) | 37.9 (11.8) | 36.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 70 | 70 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/white | 27 | 25 | 52
  African American/black | 27 | 25 | 52
  Native American | 1 | 3 | 4
  Asian/Pacific Islander | 2 | 1 | 3
  Hispanic/Latino | 11 | 14 | 25
  Multiracial/Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Time From Exposure to Truvada Initiation
Description: Time to initiation is defined as the number of hours between exposure to viral inoculum and initiation of the Truvada medication regimen.
Time Frame: 6-month follow-up
Population: 40 participants with evaluable data initiated Truvada during the course of the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Contingency Management | Yoked Contingency Management
Number analyzed (Participants) | 26 | 14
hours | 32.8 (15.1) | 33.0 (16.1)

2. Secondary Outcome: Abstinence From Stimulant Drug Use (Cocaine, Amphetamine, Methamphetamine)
Description: Abstinence will be measured using thrice weekly urine drug screens and self-report
Time Frame: Thrice-weekly for 8 weeks
Population: 170 participants enrolled in the study, of which 30 were involved in a protocol violation that rendered their data un-analyzable. The final analytical sample is N = 140.
Measure: Mean (Standard Deviation); unit: Stimulant-free urinalyses
Arm/Group | Contingency Management | Yoked Contingency Management
Number analyzed (Participants) | 70 | 70
Stimulant-free urinalyses | 8.9 (9.2) | 6.0 (6.1)

3. Primary Outcome: Medication Adherence
Description: Adherence to Truvada medication (if initiated) as assessed by self-report and pill count.
Time Frame: Daily throughout medication course
Population: 40 participants initiated Truvada, of which 30 had evaluable medication adherence and course completion data (the 10 others were involved in the protocol violation).
Measure: Number; unit: proportion
Arm/Group | Contingency Management | Yoked Contingency Management
Number analyzed (Participants) | 17 | 13
proportion | 0.75 (NA) | 0.45 (NA)

4. Primary Outcome: Course Completion
Description: PEP course completion is a dichotomous variable (0 = Not completed; 1 = Completed) that indicates whether the participant maintained sufficient adherence to the Truvada regimen to receive all 28 doses of the medication. Note: Missing 3 Truvada doses in a row terminated the PEP-intervention and prevented Course Completion.
Time Frame: 28-days post initiation
Population: 40 participants initiated PEP during the study, of which 30 had evaluable course completion data.
Measure: Number; unit: participants
Arm/Group | Contingency Management | Yoked Contingency Management
Number analyzed (Participants) | 17 | 13
participants | 12 | 4

ADVERSE EVENTS:
Time Frame: From enrollment to 6-month follow-up.
Arm/Group | Contingency Management | Yoked Contingency Management
Serious Adverse Events (participants affected / at risk) | 1/70 | 1/70
Other Adverse Events (participants affected / at risk) | 8/70 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contingency Management (N=70) | Yoked Contingency Management (N=70)
Suicidal Ideation/Exacerbated Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Participant was hospitalized for suicidality. He was held in the emergency department overnight, and was subsequently transferred from the emergency room to another hospital for treatment of suicidal ideation.
Death (General disorders) | 0 (0) | 1 (1) — Participant died of acute heroin overdose. Not study related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contingency Management (N=70) | Yoked Contingency Management (N=70)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcer on Hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Painless
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tooth Pain (General disorders) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0)
Throat Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hot Flashes (General disorders) | 1 (1) | 0 (0)
Profuse Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No